CLINICAL TRIAL: NCT05427526
Title: Outcome of Zeiss AT LARA EDOF Lens Implantation in Vitrectomized Eyes
Acronym: LARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: S65356
Record Dates: First submitted 2022-01-26; First posted 2022-06-22 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Vitreous Disorder; Cataract
Keywords: LARA EDOF lens; Intra ocular lensimplantation; cataract; vitrectomy
MeSH Terms: conditions — Cataract | interventions — Lens Implantation, Intraocular

STUDY DESIGN:
Intervention Model Description: group 1: patients that had a LARA IOL implanted in combination with vitrectomy group 2: patients that had a LARA IOL implanted in during surgery for cataract secondary to vitrectomy
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: LARA IOL implanted in combination with vitrectomy. (Active Comparator): intraocular lens implantation in combination with vitrectomy
  Interventions: Procedure: intraocular lens implantation
- group 2: LARA IOL implanted in during surgery for cataract secondary to vitrectomy (Active Comparator): intraocular lens implantation during surgery for cataract secondary to vitrectomy
  Interventions: Procedure: intraocular lens implantation

INTERVENTIONS:
Procedure: intraocular lens implantation — Lens surgery during or before vitrectomy surgery.

SUMMARY:
To determine the surgical outcome and patient satisfaction in patients who underwent AT LARA lens implantation during or after vitrectomy at a relatively young age (around 55 years of age), mostly to treat (urgent) retinal detachment.

DETAILED DESCRIPTION:
The surgical outcome is defined as the patient satisfaction determined by patient questionnaires.

* Visual quality: CatQuest questionnaire
* Near vision: NAVS questionnaire
* Glare: APPLES questionnaire

These questionnaires are standardized and validated, although no cut-off values have been determined. Hence, the results drawn from these questionnaires are descriptive only.

ELIGIBILITY:
Inclusion Criteria:

* patients that had a LARA IOL implanted in combination with vitrectomy.
* patients that had a LARA IOL implanted in during surgery for cataract secondary to vitrectomy.

Exclusion Criteria:

* Patients with a LARA IOL implanted without concomitant or earlier vitrectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
visual quality | 2 weeks
  Catquest questionnaire measuring activity limitations in daily life due to poor vision
near vision | 2 weeks
  Near Activity Visual Questionnaire (NAVQ) evaluating the near vision
glare | 2 weeks
  The Assessment of Photic Phenomena and Lens Effects (APPLES) questionnaire assessing the glare

SECONDARY OUTCOMES:
Binocular performance | 2 weeks
  visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No